CLINICAL TRIAL: NCT03228719
Title: A Novel Physical Therapy Administered Physical Activity Intervention After TKR: A Randomized Control Trial
Brief Title: A Physical Therapist Administered Physical Activity Intervention After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Daniel K. White, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 946165-97
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity
Keywords: Total Knee Replacement; Physical Therapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Standardized Outpatient Physical Therapy after TKR
  Interventions: Other: Standardized PT after TKR
- Intervention Group (Experimental): Standardized Outpatient Physical Therapy after TKR with a Physical Activity Intervention
  Interventions: Behavioral: Standardize PT after TKR with a Physical Activity Intervention; Other: Standardized PT after TKR

INTERVENTIONS:
Behavioral: Standardize PT after TKR with a Physical Activity Intervention — Standardized PT and a physical activity intervention. Participants will be provided a FitbitTM Zip within one week after enrolling in the study. Participants will self-track their steps/day using their FitbitTM Zip. Participants ≤ 3 weeks' post-operative TKR are expected to maintain and not increase steps/day. Beyond 3 weeks after surgery, step goals will be initiated and evaluated on a weekly basis. Progression of weekly steps/day goal will be a joint decision between the participant and physical therapist. As a guide, a 10-20% increase in steps/day until at least 6,000 steps/day is achieved. Each week the physical therapist will review the participant's steps/day goal and if at least 4 of the 7 previous days per week were at or above the prior week's steps/day goal, then next week's steps/day goal will increase. The physical therapist will discuss current steps/day with the participant using the Fitbit TM Zip and set a personalized steps/day goal each week during PT.
  Arms: Intervention Group
Other: Standardized PT after TKR — Participants in the control group will receive standardized PT provided by a licensed physical therapist at UDPT using the University of Delaware's Rehabilitation Guidelines for Unilateral Total Knee Replacement. Standardized PT also includes a printed home exercise program with an exercise log that is updated weekly by a physical therapist. PT appointment times range from 45-60 minutes with appointment occurring 1-3 times a week for 6-8 weeks.

SUMMARY:
Background: The definitive treatment for knee osteoarthritis is Total Knee Replacement (TKR), which results in clinically meaningful improvements in pain and physical function. However, evidence suggests that physical activity remains unchanged after TKR. This randomized clinical trial is investigating the efficacy, fidelity, and safety of a physical therapist administered physical activity intervention for people after TKR.

Methods/Design: One hundred and twenty individuals, over the age of 45, who seek outpatient Physical Therapy (PT) following a unilateral TKR will be randomized into a control and intervention group. The intervention group will receive a weekly physical activity intervention during PT, which includes a FitbitTM monitor, individualized step goals, and face-to-face feedback provided by the physical therapist. Efficacy of the intervention will be measured by minutes/week spent in Moderate-to-Vigorous Physical Activity (MPVA) using an Actigraph GT3X monitor from enrollment to discharge, 6 months and 12 months from discharge from PT. The association of self-efficacy for exercise and kinesiophobia with physical activity will also be measured at the same time points. Fidelity and safety of the intervention will be assessed during outpatient PT.

Discussion: This study is designed to fill a critical clinical need to increase physical activity after TKR. The primary objective of the study is to evaluate the efficacy of a physical therapist administered physical activity intervention for people after TKR. The secondary objectives are to evaluate the fidelity and safety of a physical therapist administered physical activity intervention for people after TKR and to investigate changes in self-reported and performance-based physical function after a physical therapist administered physical activity intervention for people after TKR. The tertiary objective is to explore the association of psychosocial factors with physical activity 6 and 12 months after discharge from a physical therapist administered physical activity intervention for people after TKR. The findings will be used to support a large multi-site clinical trial to test the effectiveness, implementation, and cost of this intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 45
2. Seeking outpatient physical therapy for a unilateral TKR

Exclusion Criteria:

1. Not interested in increasing physical activity
2. Any other medical conditions that limit your physical activity
3. Have had or are planning on having another leg surgery within 6 months that is unrelated to your TKR surgery
4. Previously enrolled in a physical activity intervention study at this clinic

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K White, PT, ScD, MSc, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christiansen MB, Thoma LM, Master H, Schmitt LA, Pohlig R, White DK. A Physical Therapist-Administered Physical Activity Intervention After Total Knee Replacement: Protocol for a Randomized Controlled Trial. Phys Ther. 2018 Jul 1;98(7):578-584. doi: 10.1093/ptj/pzy037. PMID 29608733

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study protocol enrolled n=125 study participants, however prior to randomization n=5 subjects dropped out of the study. Hence, n=120 study participants were randomized, which is the number stated in the participant flow module.
Groups:
- Control Group: Standardized Outpatient Physical Therapy after Total Knee Replacement
- Intervention Group: Standardized Outpatient Physical Therapy after Total Knee Replacement with a Physical Activity Intervention
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 58 | 62
Completed | 54 | 56
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Population: This is the analytic sample size that included
  * All subjects who were randomized
  * The ActiGraph monitor was worn for > 4 days of 10 hours of wear at baseline.
Groups:
- Intervention: Group received Outpatient Physical Therapy Plus a Physical Activity Intervention
- Control: Group received Outpatient Physical Therapy only
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.80 (8.65) | 64.70 (6.57) | 66.30 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 59
  Male | 23 | 28 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 54 | 55 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 54 | 52 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110
Moderate to Vigorous Intensity Physical Activity [Mean (Standard Deviation); unit: Minutes/day] | 3.94 (9.12) | 6.70 (9.04) | 5.32 (9.15)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Measured by an Actigraph GT3X Monitor
Description: Time spent in Moderate to Vigorous Physical Activity (MVPA) average minutes/week
Time Frame: Baseline, discharge from PT, and 6 months after PT discharge
Measure: Median (Inter-Quartile Range); unit: Minutes/Week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 55 | 55
Minutes/Week
  Baseline MVPA | 9.8 [4.2 to 15.4] | 23.8 [11.2 to 36.4]
  Discharge MVPA | 63 [35 to 91] | 86.8 [48.3 to 125.3]
  6 Months MVPA | 55.3 [15.4 to 95.2] | 89.6 [31.5 to 147.74]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from enrollment until the last follow up, i.e., at 12 months after discharge from outpatient physical therapy, up to 16 months.
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/62
Serious Adverse Events (participants affected / at risk) | 9/58 | 5/62
Other Adverse Events (participants affected / at risk) | 29/58 | 39/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=58) | Intervention Group (N=62)
Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Surgical Complication (Surgical and medical procedures) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cancer Diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Knee Replacement Revision (Surgical and medical procedures) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=58) | Intervention Group (N=62)
DVT (Vascular disorders) | 5 (5) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (10)
Pain (Musculoskeletal and connective tissue disorders) | 22 (22) | 35 (35)
Swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT03228719/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT03228719/SAP_005.pdf
  • Informed Consent Form (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03228719/ICF_002.pdf